CLINICAL TRIAL: NCT03605264
Title: Biomarkers Neutrophil Gelatinase Associated Lipocalin, Interleukin 18 as Predictors of Acute Kidney Injury in Renal Transplant Recipients A Pilot Study
Brief Title: Biomarkers NGAL, IL 18 as Predictors of Acute Kidney Injury in Renal Transplant Recipients
Status: Completed | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-Renal Biomarkers-1
Record Dates: First submitted 2018-07-20; First posted 2018-07-30 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2018-08

CONDITIONS: Kidney Transplant; Complications; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples collected in Ethylenediaminetetraacetic Acid(EDTA) vials
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Slow Graft Function: Slow Graft function(SGF) is defined as a failure of serum creatinine to fall by 70% at postoperative day 7 after renal transplantation.
- Immediate Graft Function: Immediate graft function(IGF) is defined as a fall of serum creatinine of 70% at postoperative day 7 after renal transplantation.

SUMMARY:
New markers of AKI including plasma Neutrophil Gelatinase Associated Lipocalin (NGAL) and Interleukin 18(IL-18) may form a biomarker panel that may help predict AKI earlier in the course of disease than creatinine.

Biomarkers for renal injury decreases following successful Renal transplantation. The level of decrease in biomarkers, correlates with the renal graft function, and this fall occurs earlier than the fall in creatinine and/or increase in the Urine output. Should graft dysfunction occurs, investigating the fall in biomarkers could provide a window of opportunity for therapeutic interventions and also guide in evaluating the effectiveness of such interventions. NGAL is a 25 kilo Dalton(kDa) ligand-binding protein of the lipocalin family, present in human tissues including kidney. NGAL is induced early in ischemic or nephrotoxic injury to the kidney. It has also been evaluated as a biomarker of acute injury in kidney transplantation. Interleukin (IL)-18 is synthesized as an inactive 23 kDa precursor by several tissues including monocytes, macrophages, and proximal tubular epithelial cells. Urine IL-18 is elevated in patients with acute tubular necrosis and in urinary tract infection, chronic renal insufficiency, and prerenal azotemia.

Delayed graft function and slow graft function are associated with poor graft survival at one year. Early prediction of graft dysfunction could help prognosticate and initiate renoprotective measures. Urine biomarkers including NGAL and IL 18 have shown promise in this regard, but it may be fraught with risk of biomarker dilution, an effect of urinary flow rate on biomarker levels. The investigators hypothesized that plasma NGAL and plasma IL-18 can detect reduced renal graft function in renal transplant recipients within the first 2 postoperative days.

DETAILED DESCRIPTION:
Creatinine is widely used as a marker of kidney function. The use of Creatinine has many confounding factors, and it rises only after loss of 50% of renal function. This time lost in rise of serum creatinine gives rise to the risk of missing time window that may be used to prevent progress of Acute Kidney Injury (AKI).

NGAL and IL 18 are a panel of new biomarkers associated with acute kidney injury, and their levels correlate with an improvement of graft function in renal transplant recipients. Precise and early detection of a failing graft can prompt multiple investigations and interventions which may ultimately aid in maintaining the graft.

The serum levels were measured to avoid the dilution effect and output variability of urine samples.

The investigators measure the serum NGAL and IL-18 for the first 2 post-operative days after renal transplantation, and check if the trends correlate with long term graft survival and function.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing renal transplant surgery

Exclusion Criteria:

* Patients with sepsis
* Patients diagnosed with malignancy
* Patients on immunosuppressants for other indications
* Denial to participation
* Patients undergoing re-transplantation
* Pregnant Women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is patients undergoing renal transplantation
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-01-15 (Actual); Study Completion 2017-02-15 (Actual)

PRIMARY OUTCOMES:
Slow Graft Function | 7 days
  failure of serum creatinine to fall by 70% at postoperative day 7 after renal transplantation.
Early Graft Loss(EGL) | 30 days
  Early Graft Loss was defined as graft nephrectomy or loss of kidney transplant function resulting in the recipient becoming dialysis dependent within 30 days of kidney transplantation (and never achieving graft function thereafter) or death with a non-functioning graft within 30 days